CLINICAL TRIAL: NCT06622083
Title: Effect of Single Session Aerobic Exercise on Learning Outcomes of Students in Practical Courses: A Randomized Controlled Trial
Brief Title: Effect of Aerobic Exercise on Learning Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Responsible Party: Principal Investigator, Seda Yakit Yesilyurt, Assistant Prof., Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SYY 4
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-10

CONDITIONS: Learning Outcome; Pelvic Floor; Student; Education; Aerobic Exercises; Physiotherapy and Rehabilitation
MeSH Terms: interventions — Educational Status; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education group (Active Comparator): Participants in this group will receive 40 minutes of both theoretical and practical education.
  Interventions: Other: Education
- Education and Aerobic exercise group (Experimental): Participants in the exercise group will undergo an aerobic exercise program Following the exercise, participants will receive 40 minutes of both theoretical and practical education.
  Interventions: Other: Education and Aerobic exercise

INTERVENTIONS:
Other: Education — Students in both groups will be given 40 minutes of both theoretical and practical training on the anatomy of the pelvic floor, its contraction mechanism, function and dysfunctions, evaluation and physiotherapy and rehabilitation. Theoretical training will be given through presentation and question-answer techniques containing this information, and practical training will be given through a pelvic model and gynecological examination simulator.
  Arms: Education group
Other: Education and Aerobic exercise — Participants in the exercise group will undergo an aerobic exercise program using the Monark 938E Nova Ergometer and software before the training session. The bike operates with its computer software integrated with the ECG system. The aerobic exercise program will consist of 3-5 minutes of warm-up, 20 minutes of exercise, and 3-5 minutes of cool-down, performed at a moderate intensity. During the exercise session, heart rate will be recorded every 5 minutes using a Polar ECG sensor connected via Bluetooth to the 938E Nova Ergometer, while perceived exertion will be measured using Borg's 6-20 rating scale
  Arms: Education and Aerobic exercise group

SUMMARY:
Most studies have reported that physical activity positively affects memory, observation, problem-solving, decision-making, and specific skills (e.g., reading and mathematics). From an acute perspective, a single exercise session performed before, during, and after a learning task has been shown to improve various memory and executive functions (e.g., decision-making, goal planning, task switching). A meta-analysis indicated that exercise performed close to learning tasks enhances short-term memory (e.g., information that disappears within a few seconds) and long-term memory (e.g., information recalled after long time delays). Practical training is necessary in physiotherapy education programs. Practical training includes laboratory work at school, profession-related projects, and clinical internships. Practical work learning prepares students for their profession, job roles, and professional identity. Furthermore, increasing practical applications, such as assessment and practice on models, will also enhance problem-based learning. Therefore, new approaches that enhance learning in practical training in the field of physiotherapy and rehabilitation may contribute to the development of knowledgeable and qualified physiotherapists.

In this context, this study was designed to evaluate the effect of a single session of aerobic exercise before a lecture on pelvic floor rehabilitation, which includes practical methods, on the learning outcomes of the course.

ELIGIBILITY:
Inclusion Criteria:

* Being a Physiotherapy and Rehabilitation student
* Not having taken a course/training on pelvic floor rehabilitation,
* Being between the ages of 18-22,
* Being a volunteer,
* Being literate in Turkish.

Exclusion criteria:

* Those with a high metabolic aerobic threshold according to the International Physical Activity Questionnaire (3000 METs and above),
* Students who answered "Yes" to any of the 7 questions in the General Health Questions section of the Exercise Readiness for All Questionnaire,
* Those with a history of neurological disease or epilepsy,
* Those with problems that prevent participation in exercise such as hypertension or other cardiovascular diseases.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Change in Pelvic Floor Health Knowledge Test score | 1 week after the intervention
  The Pelvic Floor Health Knowledge Test (PFHKT) will be used to assess the pelvic floor knowledge level of the students participating in the study. The PFHKT was developed by Çelenay Toprak, and its Turkish validity was assessed through face validity, content validity, and construct validity analyses. The PFHKT, designed to measure participants; knowledge of pelvic floor health, consists of 29 items. The test uses a dichotomous scoring system where correct answers are scored as 1; and incorrect or unknown answers are scored 0. The minimum score is 0; and the maximum score is 29. As the score increases, the individuals knowledge of pelvic floor health also increases.
Change in Pelvic Floor Health Knowledge Test score | after the intervention
  The Pelvic Floor Health Knowledge Test (PFHKT) will be used to assess the pelvic floor knowledge level of the students participating in the study. The PFHKT was developed by Çelenay Toprak, and its Turkish validity was assessed through face validity, content validity, and construct validity analyses. The PFHKT, designed to measure participants; knowledge of pelvic floor health, consists of 29 items. The test uses a dichotomous scoring system where correct answers are scored as 1; and incorrect or unknown answers are scored 0. The minimum score is 0; and the maximum score is 29. As the score increases, the individuals knowledge of pelvic floor health also increases.

SECONDARY OUTCOMES:
Evaluation of 10 points determined on the pelvis model | at baseline
  Ten points will be marked on the pelvic model, and participants will be asked to correctly write the specified points.
Evaluation of 10 points determined on the pelvis model | after the intervention
  Ten points will be marked on the pelvic model, and participants will be asked to correctly write the specified points.
Evaluation of 10 points determined on the pelvis model | 1 week after the intervention
  Ten points will be marked on the pelvic model, and participants will be asked to correctly write the specified points.
Evaluation of digital palpation on the model | at baseline
  Digital palpation will be evaluated on the gynecological examination simulator (Can and Cannot Apply).
Evaluation of digital palpation on the model | after the intervention
  Digital palpation will be evaluated on the gynecological examination simulator (Can and Cannot Apply).
Evaluation of digital palpation on the model | 1 week after the intervention
  Digital palpation will be evaluated on the gynecological examination simulator (Can and Cannot Apply).

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir University of Economics, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No